CLINICAL TRIAL: NCT02693717
Title: A Phase II Trial to Evaluate Pemetrexed Clinical Responses in Relation to Tumor MTAP Gene Status in Patients With Previously Treated Metastatic Urothelial Carcinoma
Brief Title: Pemetrexed Disodium in Treating Patients With Previously Treated Metastatic Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was closed due to the changing efficacy of treatments for metastatic urothelial cancer.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0592; NCI-2016-00390 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0592 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pemetrexed disodium) (Experimental): Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidine-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt

SUMMARY:
This phase II trial studies how well pemetrexed disodium works in treating patients with previously treated urothelial cancer that has spread from the primary site (place where it started) to other places in the body. Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the objective response rates (ORR) to pemetrexed disodium (pemetrexed) in patients with MTAP-deficient metastatic bladder cancer.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) for patients with MTAP-deficient metastatic bladder cancer treated with pemetrexed.

II. To determine the overall survival (OS) for patients with MTAP-deficient metastatic bladder cancer treated with pemetrexed.

III. Evaluate the toxicity of pemetrexed therapy for patients with MTAP-deficient metastatic bladder cancer.

IV. Collect blood, urine, and tissue for future translational studies.

OUTLINE:

Patients receive pemetrexed disodium intravenously (IV) over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 weeks and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmation of metastatic urothelial carcinoma; patients must have sufficient tumor tissues for future MTAP testing and research; histological variants such as glandular, squamous, sarcomatoid, micropapillary, plasmacytoid, and small cell changes will not be allowed for this trial unless these tumors are MTAP-deficient
* All patients must have measurable disease and tumors of sufficient sizes for biopsy; in general, liver and lung lesions should be at least 1.0 cm, and patients with lymph node-only disease should have lesions of >= 1.5 cm in shortest dimension; patients with disease confined to bone may be eligible if a measurable lytic defect is present; the study principal investigator (PI) is the final arbiter in questions related to measurability; patients with a three-dimensional mass or pelvic sidewall fixation on bladder examination under anesthesia are considered to have measurable disease
* Patients who have received any non-anti-folate containing neoadjuvant or systemic chemotherapy are eligible; any prior intravesical therapy, or immunotherapy is allowed
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 x upper limit normal (ULN), or =< 5 x ULN if documented liver metastases are present
* Total bilirubin =< 1.5 x ULN, except subjects with Gilbert's syndrome or liver metastases, who must have a baseline total bilirubin =< 3.0 mg/dL
* Absolute neutrophil count (ANC) >= 1500
* Platelets >= 100,000
* Normal serum creatinine, or a creatinine clearance >= 40 ml/min (either measured using a 24 hour urine, calculated using Cockroft-Gault, or estimated using the Modification of Diet in Renal Disease [MDRD] method from the National Kidney Disease Education Program [NKDEP] [the method reported by M D Anderson Cancer Center (MDACC) laboratories])
* Females of childbearing potential who are sexually active with a non-sterilized male partner and non-sterilized males must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 180 days after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician
* Females of childbearing potential must also refrain from egg cell donation for 180 days after the final dose of investigational product;

  * Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
  * A highly effective method of contraception is defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly; the acceptable methods of contraception are: barrier method (e.g. male condom with spermicide, copper T intrauterine device, or levonorgestrel-releasing intrauterine system - Mirena) or hormonal methods (e.g. implants, hormone shot or injection, combined pill, minipill, or patch); non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from days 1-180 post last dose; in addition, they must refrain from sperm donation for 180 days after the final dose of investigational product
* The ability to interrupt nonsteroidal antiinflammatory drug (NSAIDS) 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed
* The ability to take folic acid, vitamin B12, and dexamethasone according to protocol

Exclusion Criteria:

* Primary central nervous system (CNS) malignancies or CNS metastases, including leptomeningeal metastases, are not allowed; subjects with previously treated brain metastases will be allowed if the brain metastases have been stable for at least 3 months following prior treatment (radiotherapy or surgery)
* Patients who received previous anti-folate-containing chemotherapy
* Any other malignancy from which the patient has been disease-free for less than 3 years, except for non-melanoma skin cancer, controlled localized prostate cancer, in situ carcinoma of any site
* Women who are pregnant or breastfeeding
* Presence of third space fluid which cannot be controlled by drainage; for patients who develop or have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before or during initiation of pemetrexed therapy, consideration should be given to draining the effusion prior to dosing; however, if, in the investigator's opinion, the effusion represents progression of disease, the patient should be discontinued from study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Gao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Alhalabi O, Chen J, Zhang Y, Lu Y, Wang Q, Ramachandran S, Tidwell RS, Han G, Yan X, Meng J, Wang R, Hoang AG, Wang WL, Song J, Lopez L, Andreev-Drakhlin A, Siefker-Radtke A, Zhang X, Benedict WF, Shah AY, Wang J, Msaouel P, Zhang M, Guo CC, Czerniak B, Behrens C, Soto L, Papadimitrakopoulou V, Lewis J, Rinsurongkawong W, Rinsurongkawong V, Lee J, Roth J, Swisher S, Wistuba I, Heymach J, Wang J, Campbell MT, Efstathiou E, Titus M, Logothetis CJ, Ho TH, Zhang J, Wang L, Gao J. MTAP deficiency creates an exploitable target for antifolate therapy in 9p21-loss cancers. Nat Commun. 2022 Apr 4;13(1):1797. doi: 10.1038/s41467-022-29397-z. PMID 35379845
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were accrued starting in Sept 2017 through January 2019.
Groups:
- Pemetrexed: Intravenous infusion 500 mg/m2 every 21 days
Period: Overall Study
Arm/Group | Pemetrexed
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 73.6 [68 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates
Description: Will be defined as the number of subjects with complete response or partial response by Response Assessment in Solid Tumors 1.1 criteria divided by the total number of subjects receiving their first dose of trial therapy. Objective response rates will be summarized using descriptive statistics.
Time Frame: Up to 5 years
Population: Study terminated early, no data collected
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be estimated and plotted with the methods of Kaplan and Meier.
Time Frame: Time from trial entry to the first documented tumor progression as determined by the investigator using the Response Evaluation Criteria in Solid Tumors 1.1 criteria or death from any cause, assessed at 2 years
Population: Study terminated early, no data collected
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival will be estimated and plotted with the methods of Kaplan and Meier.
Time Frame: Time from trial entry to death from any cause, assessed at 2 years
Population: Study terminated early, no data collected
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Study terminated early, no data collected
Arm/Group | Pemetrexed
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This protocol was stopped early as it was considered unethical. A new protocol with the same study drugs plus an immune check point drug was added. There is no data to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT02693717/Prot_SAP_000.pdf